CLINICAL TRIAL: NCT02418429
Title: Combined Effects of Dietary Supplementation With Dietary Resistant Starch (RS) and Whey Protein on Resting Energy Expenditure and Blood Sugar and Insulin Responses in Lean and Obese Men and Women
Brief Title: Resistant Starch and Whey Protein on Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1307-348
Record Dates: First submitted 2015-04-07; First posted 2015-04-16 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Weight Loss
Keywords: fat oxidation; hunger; resistant starch; whey protein
MeSH Terms: conditions — Weight Loss | interventions — Whey Proteins; Resistant Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- waxy maize starch (Active Comparator): pancake test meal - waxy maize starch
  Interventions: Other: waxy maize starch
- waxy maize starch and whey protein (Active Comparator): pancake test meal - waxy maize starch and whey protein
  Interventions: Other: waxy maize starch; Other: waxy maize starch and Whey Protein
- resistant starch (Active Comparator): pancake test meal - resistant starch
  Interventions: Other: Resistant Starch
- resistant starch and whey protein (Active Comparator): pancake test meal - resistant starch and whey protein
  Interventions: Other: Resistant Starch; Other: resistant starch and whey protein

INTERVENTIONS:
Other: waxy maize starch — pancake test meal with waxy maize starch only
  Other Names: WMS
  Arms: waxy maize starch; waxy maize starch and whey protein
Other: waxy maize starch and Whey Protein — pancake test meal with waxy maize starch and whey protein
  Other Names: WMS-WP
  Arms: waxy maize starch and whey protein
Other: Resistant Starch — pancake test meal with resistant starch only
  Other Names: RS
  Arms: resistant starch; resistant starch and whey protein
Other: resistant starch and whey protein — pancake test meal with resistant starch and whey protein
  Other Names: RS-WP
  Arms: resistant starch and whey protein

SUMMARY:
Recent evidence shows that dietary supplementation with resistant starch (RS) increases fat catabolism and resting energy expenditure and decreases plasma insulin and glucose responses as well as the gut-derived hormone, glucose-dependent insulinotropic polypeptide (GIP). Consumption of whey protein has also been shown to increase energy expenditure and favorably affect gut hormones. Thus, investigators tested consumption of both RS and whey protein on energy expenditure and gut hormones in lean and obese women and men.

DETAILED DESCRIPTION:
Consumed separately, resistant starch (RS) and whey protein (WP) favorably affect energy metabolism and gut hormones, as well as suppress feelings of hunger. These findings are important because release of certain gut hormones (i.e., GIP) is associated with a lower resting energy expenditure (REE) in healthy humans. Interestingly, a recent study showed that ingestion of RS reduces postprandial GIP and increases postprandial REE and fat utilization in healthy men and therefore may be an effective strategy in weight management. Thus, there is a need to replicate these findings in a healthy cohort of lean and obese women and men.

The purpose of this study was to examine the effects of RS on the number of calories burned after eating a meal, as well as specific hormones that are released from the stomach and intestines following meal ingestion in healthy lean and obese women and men. Investigators used a single ingestion of a meal supplemented with or without the resistant starch and whey protein.

ELIGIBILITY:
Inclusion Criteria:

* overweight or lean but otherwise healthy

Exclusion Criteria:

* Participants will be excluded if they smoke; have experienced excessive weight loss/gain of > ±2kg in the previous 2 months; are currently taking medications for cardiovascular or metabolic disease.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in fat oxidation from Baseline to 180 Minutes Postprandial | time 0, 60, 120, 180 minutes
  indirect calorimetry of fuel utilization

SECONDARY OUTCOMES:
Change in gut hormones from Baseline to 180 Minutes Postprandial | time 0, 60, 120, 180 minutes
  gastro-entero-pancreatic hormones
Change in self-reported feelings of hunger, fullness, satiation from Baseline to 180 Minutes Postprandial | time 0, 60, 120, 180 minutes
  visual analog scale of hunger, fullness and satiation

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, PhD, Principal Investigator — Skidmore College

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gentile CL, Ward E, Holst JJ, Astrup A, Ormsbee MJ, Connelly S, Arciero PJ. Resistant starch and protein intake enhances fat oxidation and feelings of fullness in lean and overweight/obese women. Nutr J. 2015 Oct 29;14:113. doi: 10.1186/s12937-015-0104-2. PMID 26514213